CLINICAL TRIAL: NCT00939653
Title: T2007-002 A Phase II Study of Clofarabine With Etoposide and Cyclophosphamide in Relapsed/Refractory AML (IND 104,650)
Brief Title: T2007-002 Clofarabine, Etoposide, Cyclophosphamide in Relapsed Acute Myelogenous Leukemia (AML)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to insufficient research institution participation and patient enrollment
Sponsor: Therapeutic Advances in Childhood Leukemia Consortium (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T2007-002
Record Dates: First submitted 2009-07-13; First posted 2009-07-15 (Estimated); Results first posted 2020-02-19 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Relapsed Acute Myelogenous Leukemia
Keywords: relapsed; relapse; refractory; AML; Acute myelogenous leukemia; Relapsed AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — Clofarabine; Etoposide; etoposide phosphate; Cyclophosphamide; Filgrastim; Granulocyte Colony-Stimulating Factor; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm - Clofarabine with Chemo (Experimental): All patients receive the same treatment regimen consisting of clofarabine, etoposide, cyclophosphamide, cytarabine, and filgrastim. Up to 4 courses of therapy may be given.
  Interventions: Drug: Clofarabine; Drug: Etoposide; Drug: Cyclophosphamide; Drug: Filgrastim; Drug: Cytarabine

INTERVENTIONS:
Drug: Clofarabine — 40 mg/m2/day IV over 2 hours (given at hours 0 to 2) on days 1 through 5.
  Other Names: Clolar
Drug: Etoposide — 100 mg/m2/day IV over 2 hours (given at hours 2 to 4) on days 1 through 5.
  Other Names: VP-16; VePesid; Etopophos
Drug: Cyclophosphamide — 440 mg/m2/day IV as a 30-60 minute infusion (given at hours 4 to 5) on days 1 through 5.
  Other Names: Cytoxan
Drug: Filgrastim — Administered in Courses 1 and 2 only. 5 micrograms/kg/day IV or SC will begin on Day 6 and end when the ANC is > 1000 x 2 days.
  Other Names: Neupogen; G-CSF; GCSF; Granulocyte Colony Stimulating Factor
Drug: Cytarabine — Given intrathecally on day 1 at the dose defined by age below:
  30 mg for patients age 1-1.99 50 mg for patients age 2-2.99 70 mg for patients >3 years of age
  Other Names: Cytosine Arabinoside; Ara-C; Cytosar; AraC

SUMMARY:
Clofarabine is a drug approved by the FDA (Food and Drug Administration) for treating children (age 1-21) with leukemia. This research study will use clofarabine with two other cancer fighting drugs. Clofarabine will be used together with etoposide (VePesid®, VP-16) and cyclophosphamide (Cytoxan®).

DETAILED DESCRIPTION:
Clofarabine, etoposide and cyclophosphamide have been used together in a phase I study to find out the highest doses of these drugs that can be safely given to children with relapsed or refractory leukemia. This study is a phase II study which will use the drugs to study how well these drugs work against AML. This study will also examine the safety of this drug combination.

ELIGIBILITY:
Inclusion Criteria:

* Age: patients must be ≥ 1 and ≤ 21 years of age at the of study entry.
* Diagnosis:

  * Patients must have a diagnosis of first or second relapse or refractory acute myelogenous leukemia (AML) according to WHO classification with ≥ 5% blasts in the bone marrow, with or without extramedullary disease.
  * Patients may have CNS 1 or CNS 2 disease but not CNS 3.
* Performance Level: Karnofsky > 50% for patients > 16 years of age and Lansky > 50% for patients ≤ 16 years of age.
* Prior Therapy:

  * Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study.
  * Patient has not received more than 2 previous induction attempts. (Frontline therapy is included in this count).
  * Patients must have adequate venous access.
  * At least 1 year must have elapsed since hematopoietic stem cell transplant (HSCT) and patients must not have active GVHD.
* Reproductive Function

  * Female patients of childbearing potential must have a negative serum pregnancy test confirmed within 2 weeks prior to enrollment.
  * Female patients with infants must agree not to breastfeed their infants while on this study.
  * Male and female patients of child-bearing potential must agree to use an effective method of contraception approved by the investigator during the study and for a minimum of 6 months after study treatment.
* Renal and Hepatic Function:

Patient must have adequate renal and hepatic functions as indicated by the following laboratory values:

* Patients must have a normal calculated creatinine clearance.

  * Pediatric Population (age <18): Calculated creatinine clearance ≥ 90 ml/min/1.73m2 as calculated by the Schwartz formula for estimated glomerular filtration rate (GFR) where GFR (ml/min/1.73 m2) = k*Height (cm)/serum creatinine (mg/dl). k is a proportionality constant which varies with age and is a function of urinary creatinine excretion per unit of body size; 0.45 up to 12 months of age; 0.55 children and adolescent girls; and 0.70 adolescent boys.
  * Adult Population (age ≥18): Serum creatinine ≤1.0 mg/dL; if serum creatinine >1.0 mg/dL, then the estimated glomerular filtration rate (GFR) must be >60 mL/min/1.73 m2 as calculated by the Modification of Diet in Renal Disease equation where Predicted GFR (ml/min/1.73 m2) = 186 x (Serum Creatinine)-1.154 x (age in years)-0.023 x (0.742 if patient is female) x (1.212 if patient is black.
* Total bilirubin <1.5 x ULN for age and conjugated/direct serum bilirubin ≤ ULN for age if total bilirubin is elevated.
* Aspartate transaminase (AST)/alanine transaminase (ALT) ≤ 2.5 × ULN.
* Alkaline phosphatase ≤ 2.5 × ULN.

Exclusion Criteria:

* Patients with Down Syndrome.
* Prior treatment with Clofarabine.
* Previous history of veno-occlusive disease (VOD) or findings consistent with a diagnosis of VOD, defined as: conjugated serum bilirubin > 1.4 mg/dL AND unexplained weight gain greater than 10% of baseline weight or ascites AND hepatomegaly or right upper quadrant pain without another explanation, OR reversal of portal vein flow on ultrasound, OR pathological confirmation of VOD on liver biopsy.
* Patients who have a history of cirrhosis of the liver or who are positive for hepatitis B core antibody (anti-HBc) or have a positive test for hepatitis C antibody (anti-HCV).
* Patient has received TBI.
* If it has been less than 1 year since the patient had a HSCT.
* Infection Criteria

  * Patients with a systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment).
  * Positive blood culture within 48 hours of study registration.
  * Patient required supplemental oxygen or vasopressors within 48 hours of study (Oxygen after anesthesia for procedures is ok).
* Patient is receiving or plans to receive concomitant chemotherapy, radiation therapy, or immunotherapy other than as specified in the protocol.
* Use of investigational agents within 30 days or any anticancer therapy within 2 weeks before planned drug initiation with the exception of hydroxyurea or intrathecal therapy given with the diagnostic lumbar puncture.
* Have any other severe concurrent disease, or have a history of serious organ dysfunction or disease involving the heart, kidney, liver, or other organ system that may place the patient at undue risk to undergo treatment.
* Pregnant or lactating patients.
* Any significant concurrent disease, illness, psychiatric disorder or social issue that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results.
* Have had a diagnosis of another malignancy, unless the patient has been disease-free for at least 3 years following the completion of curative intent therapy with the following exceptions:

  * Patients with treated non-melanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia, regardless of the disease-free duration, are eligible for this study if definitive treatment for the condition has been completed.
  * Patients with organ-confined prostate cancer with no evidence of recurrent or progressive disease based on prostate-specific antigen (PSA) values are also eligible for this study if hormonal therapy has been initiated or a radical prostatectomy has been performed.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2009-07-10; Primary Completion 2011-07-15 (Actual); Study Completion 2011-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Gaynon, MD, Study Chair — Children's Hospital Los Angeles; Nobuko Hijiya, MD, Study Chair — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (4):
- United States (4):
  - Childrens Hospital Los Angeles, Los Angeles, California
  - University of Miami Cancer Center, Miami, Florida
  - Children's Memorial, Chicago, Illinois
  - Childrens Hospital & Clinics of Minnesota, Minneapolis, Minnesota

REFERENCES:
- See also: For more information about this and other clinical trials, please visit the TACL website. — http://www.tacl.us

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm - Protocol Chemo Regimen: All patients receive the same treatment regimen consisting of clofarabine, etoposide, cyclophosphamide, cytarabine, and filgrastim.
  clofarabine: 40 mg/m2/day IV over 2 hours (given at hours 0 to 2) on days 1 through 5.
  etoposide: 100 mg/m2/day IV over 2 hours (given at hours 2 to 4) on days 1 through 5.
  cyclophosphamide: 440 mg/m2/day IV as a 30-60 minute infusion (given at hours 4 to 5) on days 1 through 5.
  filgrastim: 5 micrograms/kg/day IV or SC will begin on Day 6 and end when the ANC is > 1000 x 2 days.
  cytarabine: Given intrathecally on day 1 at the dose defined by age below. 30 mg for patients age 1-1.99 50 mg for patients age 2-2.99 70 mg for patients >3 years of age
Period: Treatment Course 1
Arm/Group | Single Arm - Protocol Chemo Regimen
Started | 6
Completed | 6
Not Completed | 0
Period: Treatment Course 2
Arm/Group | Single Arm - Protocol Chemo Regimen
Started (Required for all patients who achieve Complete Remission (CR) or CRp, unless proceeding to HSCT) | 2
Completed | 2
Not Completed | 0
Period: Treatment Course 3
Arm/Group | Single Arm - Protocol Chemo Regimen
Started (Patients with CR or CRp and meeting other protocol-defined criteria may proceed to Courses 3 and 4.) | 0
Completed | 0
Not Completed | 0
Period: Treatment Course 4
Arm/Group | Single Arm - Protocol Chemo Regimen
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Enrolled Patients: Baseline measures were collected for all enrolled patients.
Arm/Group | Enrolled Patients
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 1
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Achievement of Complete Remission (CR) at Reinduction
Description: Disease response assessed after chemotherapy from bone marrow aspirates/biopsies and complete blood count.
Time Frame: Between Days 22-36 or on Day 43 and weekly thereafter if peripheral counts haven't recovered
Population: Patients that completed at least 1 treatment course of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Enrolled Patients: All patient that completed at least 1 treatment course.
Arm/Group | Enrolled Patients
Number analyzed (Participants) | 6
Participants | 1

2. Primary Outcome: Death
Description: Number of participants who died.
Time Frame: From the first dose of study therapy until 30 days after last therapy dose
Measure: Count of Participants; unit: Participants
Groups:
- Enrolled Patients: All patients enrolled onto study.
Arm/Group | Enrolled Patients
Number analyzed (Participants) | 6
Participants | 4

ADVERSE EVENTS:
Time Frame: From the time of treatment start until 30 days after the last dose of protocol therapy. Specific period of time varies depending on # of courses and conditions for starting next course; collection timeframe is roughly between Days 0 and Day 150.
Description: The definition of adverse event and SAE used for data collection does not differ from that in the clinicaltrials.gov Definitions.
  Patients were evaluated regularly by the treating physician.
Arm/Group | Enrolled Patients
All-Cause Mortality (participants affected / at risk) | 4/6
Serious Adverse Events (participants affected / at risk) | 6/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enrolled Patients (N=6)
Capillary leak syndrome (Vascular disorders) | 1
Renal failure NOS (Renal and urinary disorders) | 2
Febrile Neutropenia (Blood and lymphatic system disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Grade 3 Infection (blood) (Infections and infestations) | 2
Syncope (Nervous system disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 1
Platelet count decreased (Blood and lymphatic system disorders) | 1
Hypotension NOS (Vascular disorders) | 1
Neutrophil Count (Blood and lymphatic system disorders) | 1
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension NOS (Vascular disorders) | 1
Pulmonary - Other (Respiratory, thoracic and mediastinal disorders) | 1 — Respiratory failure
Multi-organ failure (General disorders) | 1 — Infection of underlying immune suppression related to leukemia
Clostridial infection NOS (Infections and infestations) | 1 — C. Difficile, stool
Grade 4 Infection (Infections and infestations) | 2
Grade 4 ANC (Infections and infestations) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enrolled Patients (N=6)
aPTT prolonged (Investigations) | 2
Alanine aminotransferase increased (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 1
Anxiety (Psychiatric disorders) | 1
AST increased (Investigations) | 3
Blood amylase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 2
Blood creatinine increased (Investigations) | 1
Blood/Bone Marrow-Other (Blood and lymphatic system disorders) | 2 — Low Hgb, neutropenia
Constipation (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Depression (Psychiatric disorders) | 1
Dermatitis exfoliative NOS (Skin and subcutaneous tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Electrocardiogram QT prolonged (Cardiac disorders) | 1
Epistaxis (Vascular disorders) | 2
GGT increased (Investigations) | 1
Hematoma (Vascular disorders) | 1
Hemoglobin - low (Blood and lymphatic system disorders) | 4
Hemorrhagic stroke (Vascular disorders) | 1
Hyperglycemia NOS (Metabolism and nutrition disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypertension NOS (Vascular disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 4
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypoglycemia NOS (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Hypotension NOS (Vascular disorders) | 2
Infection w/ Gr 3/4 ANC (Infections and infestations) | 5 — 4 participants: blood, 1 participant: nose
Infection w/ norm ANC, Blood (Infections and infestations) | 1
Infection w/ unk ANC, Mucosa (Infections and infestations) | 1
Left ventricular failure (Cardiac disorders) | 2
Leukopenia NOS (Blood and lymphatic system disorders) | 5
Lymphopenia (Blood and lymphatic system disorders) | 1
Mouth hemorrhage (Vascular disorders) | 1
Neutrophil count (Blood and lymphatic system disorders) | 3
Pain - other (General disorders) | 1
Platelet count decreased (Blood and lymphatic system disorders) | 5
Pruritis (Skin and subcutaneous tissue disorders) | 3
Psychosis aggravated (Psychiatric disorders) | 1
Pyrexia (General disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Stomatitis (Gastrointestinal disorders) | 2
Urticaria NOS (Skin and subcutaneous tissue disorders) | 1
Vomiting NOS (Gastrointestinal disorders) | 1

LIMITATIONS AND CAVEATS:
Trial was terminated early due to loss of funding and concern that accrual goals could not be met. All six patients enrolled were deemed evaluable toxicity. No analysis was conducted on the study outcome variables.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days